CLINICAL TRIAL: NCT00012714
Title: Evaluation of Subacute Rehabilitative Care
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIR 94-125
Record Dates: First submitted 2001-03-14; First posted 2001-03-16 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2007-02

CONDITIONS: Rehabilitative Services

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Behavioral: Case management services

INTERVENTIONS:
Behavioral: Case management services

SUMMARY:
Prior rehabilitation outcome studies had many weaknesses. They had: a) evaluated rehabilitation effects only in isolated subgroups, b) focused on functional ability rather than on quality of life, c) not used randomized control groups, and d) had inadequate sample sizes. Differences in methodological approaches have resulted in inconsistent findings. The lack of long-term benefits suggests that services may need to be continued at home or in subacute care settings to optimize their effectiveness. Unfortunately, prior research did not include behavioral outcomes. The potential benefits of rehabilitative care could thus not be evaluated by these studies in more meaningful detail, and they did not accurately reflect the psychosocial objectives of rehabilitation.

DETAILED DESCRIPTION:
Background:

Prior rehabilitation outcome studies had many weaknesses. They had: a) evaluated rehabilitation effects only in isolated subgroups, b) focused on functional ability rather than on quality of life, c) not used randomized control groups, and d) had inadequate sample sizes. Differences in methodological approaches have resulted in inconsistent findings. The lack of long-term benefits suggests that services may need to be continued at home or in subacute care settings to optimize their effectiveness. Unfortunately, prior research did not include behavioral outcomes. The potential benefits of rehabilitative care could thus not be evaluated by these studies in more meaningful detail, and they did not accurately reflect the psychosocial objectives of rehabilitation.

Objectives:

The goal of this study was to measure the additive effect of outpatient, subacute rehabilitation as follow-up services to acute, inpatient rehabilitation on adults diagnosed with a disabling disorder in four major diagnostic groups (nervous, circulatory, musculoskeletal, and injury).

Methods:

A randomized clinical trial was conducted to determine the effects of subacute rehabilitative care on: 1) physical function, 2) health and mental health, 3) mortality, 4) family function, 5) personal adjustment, and 6) use of health care resources. Patients hospitalized for the first time with a disabling condition [n=180] were provided inpatient rehabilitation and then randomly assigned to either subacute rehabilitation at home [n=90] or to usual outpatient follow-up [n=90] in which only medical services were provided but no scheduled rehabilitative therapies were offered. To compare the two groups, analysis of covariance was conducted for the outcome variables. The between subjects factor was subacute rehabilitative care versus usual medical services as an outpatient.

Status:

Complete.

ELIGIBILITY:
Inclusion Criteria:

Presence of physical limitation and need for rehabilitative care as indicated by a score >1 (not independent) on the Nursing Ward Classification index; availability of a family member selected by the patient; Major Diagnostic Code (MDC) 1, 5, 8, or 21 (comprising 87% of cases)

Exclusion Criteria:

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Study Completion 2000-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald L. Evans, MSW, Principal Investigator — VA Puget Sound Health Care System Seattle Division, Seattle, WA
Locations (1):
- VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington, United States

REFERENCES:
- [Result] Evans RL, Connis RT, Haselkorn JK. Hospital-based rehabilitative care versus outpatient services: effect on functioning and health status. Disabil Rehabil. 1998 Aug;20(8):298-307. doi: 10.3109/09638289809166085. PMID 9651688
- [Result] Evans RL. Perceived functional health of disabled elderly persons in a follow-up program for primary care. Psychol Rep. 1999 Apr;84(2):553-7. doi: 10.2466/pr0.1999.84.2.553. PMID 10335067